CLINICAL TRIAL: NCT07073755
Title: A Real-World Observational Study on Post-Resistance Treatment Outcomes in Advanced Breast Cancer Patients After CDK4/6 Inhibitors, PIK3CA Inhibitors, or Trastuzumab Deruxtecan Therapy
Brief Title: Real-World Study of Post-Resistance Treatment Strategies in Advanced Breast Cancer Following CDK4/6i, PIK3CA Inhibitors, or T-DXd
Status: Recruiting | Type: Observational
Sponsor: Hunan Cancer Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: HNCA-PoReBC
Record Dates: First submitted 2025-07-09; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Metastatic Breast Cancer; Drug Resistance; Hormone Receptor-Positive Breast Cancer; HER2-positive Breast Cancer; Triple-Negative Breast Cancer (TNBC); Treatment Decisions
Keywords: Real-World Study; Treatment Resistance; Post-Progression Therapy; Metastatic Breast Cancer; Predictive Factors
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Post-Resistance Advanced Breast Cancer Patients: This cohort includes patients with advanced or metastatic breast cancer who experienced disease progression after treatment with CDK4/6 inhibitors, PIK3CA inhibitors, trastuzumab deruxtecan (T-DXd), or other targeted therapies. All patients subsequently received further systemic therapy, including chemotherapy, endocrine therapy, targeted agents, or their combinations, based on physician discretion and routine clinical practice. This observational cohort will be analyzed to assess treatment patterns, clinical outcomes (e.g., progression-free survival and overall survival), and potential prognostic or predictive factors.

SUMMARY:
This is a real-world observational study aiming to evaluate the effectiveness of post-progression treatment strategies in patients with advanced breast cancer who have developed resistance to prior targeted therapies, including CDK4/6 inhibitors, PIK3CA inhibitors, trastuzumab deruxtecan (T-DXd), or other targeted agents commonly used in clinical practice. As resistance to these therapies becomes increasingly common, optimal sequencing strategies for subsequent treatment remain unclear.

This study will collect clinical information on post-resistance systemic treatments and their outcomes, including progression-free survival, overall survival, and response rate. Baseline patient and tumor characteristics will also be collected to explore potential prognostic and predictive factors and to develop outcome prediction models that may help guide future clinical decision-making.

This is a non-interventional study based on retrospective and prospective data from routine medical care. The results are expected to provide real-world evidence to inform personalized treatment strategies for patients with advanced breast cancer following resistance to targeted therapies.

DETAILED DESCRIPTION:
Breast cancer is a heterogeneous disease, and advances in targeted therapies have significantly improved clinical outcomes, especially in hormone receptor-positive (HR+), HER2-positive, and selected triple-negative breast cancer (TNBC) subtypes. However, disease progression following treatment with targeted agents such as CDK4/6 inhibitors, PIK3CA inhibitors, and antibody-drug conjugates like trastuzumab deruxtecan (T-DXd) remains a major clinical challenge. With a growing number of post-resistance treatment options available, real-world data are urgently needed to inform evidence-based sequencing strategies in routine clinical practice.

This real-world observational study aims to investigate the treatment patterns and clinical outcomes of patients with advanced or metastatic breast cancer who experience disease progression after receiving CDK4/6 inhibitors, PIK3CA inhibitors, T-DXd, or other relevant targeted agents. The study will focus on characterizing the effectiveness of subsequent treatment regimens, including chemotherapy, endocrine therapy, additional targeted therapies, or their combinations.

In addition to evaluating clinical outcomes such as progression-free survival (PFS), overall survival (OS), objective response rate (ORR), and duration of response (DoR), the study will collect detailed baseline patient characteristics, tumor biological features, and prior treatment histories. These data will be used to identify potential prognostic and predictive factors and to develop outcome prediction models that may support personalized treatment planning in the post-resistance setting.

Patients will be identified based on medical record review, with retrospective and/or prospective data collection depending on institutional capabilities. Treatment decisions are made at the discretion of the treating physicians as part of standard clinical care. The study does not involve any experimental intervention, and no additional diagnostic or therapeutic procedures will be imposed on participants.

The ultimate goal of this study is to generate clinically relevant, real-world evidence to guide optimal treatment sequencing after resistance to targeted therapy in advanced breast cancer, and to support future clinical research and decision-making frameworks.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (≥18 years old) with histologically or cytologically confirmed advanced or metastatic breast cancer
2. Received prior treatment with at least one of the following: CDK4/6 inhibitors, PIK3CA inhibitors, trastuzumab deruxtecan (T-DXd), or other targeted therapies
3. Documented disease progression following prior targeted therapy
4. Initiated a subsequent line of systemic therapy (chemotherapy, endocrine therapy, targeted therapy, or combination) after resistance
5. Available clinical data including baseline characteristics and treatment details
6. At least one follow-up evaluation after initiation of post-resistance therapy

Exclusion Criteria:

1. Incomplete medical records or missing key clinical follow-up data
2. Concurrent diagnosis of other active malignancies (except non-melanoma skin cancer or in situ cervical cancer)
3. Known central nervous system disease requiring immediate local treatment (unless clinically stable)
4. Poor general condition with an Eastern Cooperative Oncology Group (ECOG) performance status ≥2
5. Life expectancy estimated to be less than 6 months based on clinical judgment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced breast cancer who developed resistance to targeted therapies and subsequently received systemic treatment in routine clinical practice. The study population includes diverse subtypes (HR+/HER2-, HER2+, TNBC) and reflects real-world treatment patterns in post-progression settings.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | From the start of post-resistance systemic treatment until documented disease progression or death, up to 36 months.
  Progression-Free Survival (PFS) is defined as the time from the initiation of post-progression systemic treatment (after resistance to CDK4/6 inhibitors, PIK3CA inhibitors, T-DXd, or other targeted therapies) to the date of documented disease progression or death from any cause, whichever occurs first. Disease progression will be determined based on radiological or clinical assessment, as per real-world documentation standards. Patients without progression or death at the time of analysis will be censored at the date of last follow-up.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | From start of post-resistance systemic treatment to best documented response, assessed up to 24 months.
  ORR is defined as the proportion of patients achieving a complete response (CR) or partial response (PR) to the post-progression systemic treatment, as assessed by the treating physician based on radiological or clinical documentation. Response assessment will follow real-world clinical practice without central review.
Disease Control Rate (DCR) | From treatment initiation to disease progression or last follow-up, assessed up to 24 months.
  DCR is defined as the proportion of patients who achieve complete response (CR), partial response (PR), or stable disease (SD) for at least 8 weeks after initiating post-resistance therapy. Evaluations are based on clinical or imaging assessment as documented in routine practice.
Overall Survival (OS) | From start of post-progression treatment to death or last follow-up, up to 48 months.
  OS is defined as the time from the initiation of post-resistance systemic therapy to death from any cause. Patients still alive at the time of analysis will be censored at their last known follow-up date.
Treatment-Related Adverse Events | From the start of post-resistance treatment until 30 days after treatment discontinuation, assessed up to 24 months.
  The incidence and type of treatment-related adverse events (AEs) will be collected as documented in the medical record, based on physician assessment. AEs will be classified according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0, where available.

CONTACTS AND LOCATIONS:
Locations (1):
- Hunan Cancer Hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided